CLINICAL TRIAL: NCT05548140
Title: Novel Motorized Spiral Enteroscopy Vs Single Balloon Enteroscopy In Patients With Small Bowel Disorders- A Randomized Controlled Trial
Brief Title: Novel Motorized Spiral Enteroscopy Vs Single Balloon Enteroscopy In Patients With Small Bowel Disorders- A RCT
Acronym: MOTOR-AIG-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Consultant Gastroenterologist, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MOTOR-AIG-01
Record Dates: First submitted 2022-05-25; First posted 2022-09-21 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Small Bowel Disease
Keywords: Small bowel disease; IBD; Single balloon enteroscopy; spiral enteroscopy
MeSH Terms: interventions — Single-Balloon Enteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NOVEL MOTORIZED SPIRAL ENTEROSCOPY (Experimental): This arm involves performance of spiral enteroscopy using a specialized enteroscope under general anaesthesia in patients who fulfill the inclusion criteria.
  Interventions: Device: Novel Motorized Spiral Enteroscopy
- SINGLE BALLOON ENTEROSCOPY (Active Comparator): This arm involves performance of single balloon enteroscopy using a specialized single balloon enteroscope in patients who fulfill inclusion criteria.
  Interventions: Device: Novel Motorized Spiral Enteroscopy

INTERVENTIONS:
Device: Novel Motorized Spiral Enteroscopy — This study involves performance of spiral enteroscopy in one arm and single balloon enteroscopy in the other arm in patients who satisfy inclusion criteria
  Other Names: Single Balloon Enteroscopy

SUMMARY:
STUDY OBJECTIVES:

1. Primary objective: Rate of total enteroscopy (TER) by means of NMSE or SBE with: Complete antegrade approach or combined antegrade and retrograde approach
2. Secondary objective:

   1. Technical success of anterograde and retrograde approach
   2. Procedural time (minutes)
   3. Depth of maximum insertion (cm)
   4. Diagnostic yield
   5. Therapeutic success
   6. Adverse events

DETAILED DESCRIPTION:
1. INTRODUCTION: Small-bowel (SB) disorders remain a diagnostic and therapeutic challenge for endoscopists because of its unfavourable anatomy for endoscopy. It is difficult to perform deep enteroscopy of the long redundant lengthy small intestine by the bare endoscope, most of the time operator end up in pushing the SB rather than traveling through it. Last two decades saw a paradigm shift in the management of SB disorders with the introduction of deep enteroscopy1-4, including Double-balloon enteroscopy (DBE, Fujifilm, Tokyo, Japan), Single-balloon enteroscopy5 (SBE, Olympus Medical Systems Corporation, Tokyo, Japan), and Spiral enteroscopy6 (SE, Spiral Medical, LCC, USA). The DBE and SBE techniques have had varied results as far as depth of insertion is concerned; moreover, both are time-consuming and have difficult ergonomics for the endoscopist which are a major limiting factor. Spiral enteroscopy (SE)6 was introduced in 2007, which was two-operator technique where a spiral-shaped over-tube (Discovery Small Bowel, DSB) was used to pleat the small bowel over the enteroscope by manual rotation of the over tube. Deep endoscopic access to the small bowel with all available methods is still a complex, cumbersome, time-consuming procedure, and requires high endoscopic skills. Novel Motorized Spiral Enteroscope7 (NMSE, Olympus Medical, Tokyo, Japan) is a recent advancement in the field of enteroscopy. This enteroscope works on the same principle as that of SE and comes with an integrated user controlled motor in the handle of the enteroscope. The integrated electric motor is controlled with the help of a footswitch for rotating a short spiral over tube to pleat and un-pleat the small bowel. This would increase the possibility to accelerate the procedure, facilitate insertion, and simplify the technique with a single operator. The procedure can be done both by antegrade and retrograde approaches. Data is scarce on the utility, safety and efficacy of Novel Motorized Spiral Enteroscopy (NMSE) for evaluation in patients with suspected SBD by both the routes of examination. Also there are no comparative studies between SBE and NMSE. Hence we have planned a Randomized controlled trial to compare both modalities.
2. RATIONALE: SBE is the standard procedure used for small bowel examination at our center. SBE in prior studies has shown diagnostic yield of 40-60%5 but very low TER (0-22%)4,10, with long procedure time. NMSE on the other hand has the advantage of greater TER and high diagnostic yield with shorter procedure times and minimal adverse events. Our study on NMSE11 has shown high diagnostic yield of 70%, with TER of 61% and total procedure time of around 40min. Various studies have shown the safety and efficacy of SBE and NMSE. One recent prospective study by Beyna9 et al. using NMSE for only antegrade enteroscopy showed total enteroscopy rate (TER) of 10.6% (14/132) with technical success of 97%. Majority of patients (74.2%) underwent NMSE for suspected GI bleeding. Overall diagnostic yield was 74.2% and endotherapy was done in 68.2% patients. In our study11 on NMSE, recently published, we have shown comparable technical success using both antegrade (92.85%) and retrograde (100%) routes. There was higher total enteroscopy rate of 60.6% with antegrade route showing 31.1%.This real-world scenario analysis showed that diagnostic yield of NMSE was 70% in those who successfully underwent enteroscopy and therapeutic procedures were done in almost one fourth of patients. Till date, there are no comparative data between NMSE and Balloon assisted enteroscopy techniques. Hence, we aim to compare NMSE and SBE in Randomized controlled trial.
3. STUDY METHODS / STUDY PROCEDURE / METHODS OF ASSESSMENT: Patients presenting with symptoms and signs suggestive of small bowel disorders will be admitted and investigated as per the latest guidelines2. Patients satisfying the inclusion and exclusion criteria will be randomized in one of the two arms and will undergo either NMSE or SBE. As per the presentation and indication patients in both arms will undergo antegrade or retrograde enteroscopy. Patients undergoing antegrade enteroscopy will also undergo retrograde enteroscopy if indicated in the same sitting with the aim of total enteroscopy. Patients will be managed according to the findings and will be discharged as per the conditions. Patients will be followed up in the OPD or telephonically 1 week and after 1 month of discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with small bowel disease with an indication for total enteroscopy with indeterminate imaging findings (as defined above)
2. Age > 18 years
3. Patients willing to give written consent

Exclusion Criteria:

1. Positive imaging findings (as defined)
2. Age < 18 years.
3. Contraindications for endoscopy due to comorbidities
4. Unable to provide written informed consent
5. Patients with known severe GI tract inflammation, intestinal obstruction, gastroesophageal varices that preclude a safe enteroscopy procedure
6. Coagulopathy or thrombocytopenia that couldn't be corrected by blood product transfusion
7. Pregnant patients
8. Health status American Society of Anaesthetist Classification (ASA) >3
9. Inability to tolerate sedation or general anaesthesia for any reason
10. Pediatrics patients (infants and toddlers)
11. Eosinophilic esophagitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Rate of total enteroscopy (TER) | 1 year
  Number of cases in which total small bowel examination can be performed

SECONDARY OUTCOMES:
Technical success of anterograde and retrograde approach | 1 year
  For anterograde approach, crossing of duodenal-jejunal flexure and for retrograde approach, crossing of ileo-caecal valve- describes technical success
Procedural time (minutes) | 1 year
  Time taken for the entire procedure from start to end is procedural time
Depth of maximum insertion (cm) | 1 year
  The depth till which the small bowel examination can be done. The examination can be done till we reach the expected lesion or till the scope stops further movement in small intestines
Diagnostic yield | 1 year
  Diagnostic yield is defined as the percentage of procedures that can either confirm a diagnosis from previous studies or established a new definitive diagnosis at the anatomic location identified in previous studies or findings that could explain the clinical symptoms.
Therapeutic success | 1 year
  Therapeutic success is defined as successful endoscopic interventions such as for GI bleeding, polypectomy, and so on.
Adverse events | 1 year
  Adverse events are defined as minor or major. Minor adverse event was defined as superficial esophageal or colonic trauma, sore throat less than 72 hours in duration, abdominal discomfort lasting less than 48 hours, and mild nausea or vomiting not requiring hospital admission. Major adverse events were defined as perforation, significant bleeding requiring blood products, pancreatitis, or any hospital admission related to the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Hardik Rughwani, MBBS, MD, DM, Principal Investigator — AIG Hospitals
Locations (2):
- India (2):
  - Hardik Rughwani, Hyderabad, Other
  - AIG Hospitals, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramchandani M, Rughwani H, Inavolu P, Singh AP, Tevethia HV, Jagtap N, Sekaran A, Kanakagiri H, Darishetty S, Reddy DN. Diagnostic yield and therapeutic impact of novel motorized spiral enteroscopy in small-bowel disorders: a single-center, real-world experience from a tertiary care hospital (with video). Gastrointest Endosc. 2021 Mar;93(3):616-626. doi: 10.1016/j.gie.2020.07.001. Epub 2020 Jul 12. PMID 32663489
- [Background] Rondonotti E, Spada C, Adler S, May A, Despott EJ, Koulaouzidis A, Panter S, Domagk D, Fernandez-Urien I, Rahmi G, Riccioni ME, van Hooft JE, Hassan C, Pennazio M. Small-bowel capsule endoscopy and device-assisted enteroscopy for diagnosis and treatment of small-bowel disorders: European Society of Gastrointestinal Endoscopy (ESGE) Technical Review. Endoscopy. 2018 Apr;50(4):423-446. doi: 10.1055/a-0576-0566. Epub 2018 Mar 14. PMID 29539652
- [Background] Buscaglia JM, Dunbar KB, Okolo PI 3rd, Judah J, Akerman PA, Cantero D, Draganov PV. The spiral enteroscopy training initiative: results of a prospective study evaluating the Discovery SB overtube device during small bowel enteroscopy (with video). Endoscopy. 2009 Mar;41(3):194-9. doi: 10.1055/s-0028-1119602. Epub 2009 Mar 11. PMID 19280530
- [Result] Yamamoto H, Ogata H, Matsumoto T, Ohmiya N, Ohtsuka K, Watanabe K, Yano T, Matsui T, Higuchi K, Nakamura T, Fujimoto K. Clinical Practice Guideline for Enteroscopy. Dig Endosc. 2017 Jul;29(5):519-546. doi: 10.1111/den.12883. Epub 2017 Jun 9. PMID 28370422
- See also: Clinical Practice Guideline for Enteroscopy — https://pubmed.ncbi.nlm.nih.gov/28370422/
- See also: Diagnostic yield and therapeutic impact of novel motorized spiral enteroscopy in small-bowel disorders: a single-center, real-world experience from a tertiary care hospital — https://pubmed.ncbi.nlm.nih.gov/32663489/
- See also: Small-bowel capsule endoscopy and device-assisted enteroscopy for diagnosis and treatment of small-bowel disorders: European Society of Gastrointestinal Endoscopy (ESGE) Technical Review — https://pubmed.ncbi.nlm.nih.gov/29539652/
- See also: The spiral enteroscopy training initiative: results of a prospective study evaluating the Discovery SB overtube device during small bowel enteroscopy — https://pubmed.ncbi.nlm.nih.gov/19280530/